CLINICAL TRIAL: NCT03407430
Title: A Phase II, Placebo-controlled, Double-blind, Randomized Crossover Trial of Pregabalin for the Prophylaxis of Pegfilgrastim-induced Bone Pain
Brief Title: Trial of Pregabalin for Granulocyte Colony-stimulating Factor (GCSF)-Induced Bone Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LCCC 1314
Record Dates: First submitted 2018-01-02; First posted 2018-01-23 (Actual); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Lymphoma; Pain
Keywords: Pregabalin; Bone pain; Pegfilgrastim; Supportive care; prevention
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Pain | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double blind, randomized crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin, then Placebo (Experimental): Pregabalin in cycle 1; placebo in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg twice a day (BID) for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Interventions: Drug: Pregabalin
- Placebo, then Pregabalin (Experimental): Placebo in cycle 1; pregabalin in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg BID for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — During the first chemotherapy cycle, the patient will receive pregabalin 75mg (1 capsule) BID x 4 days before pegfilgrastim 6mg subcutaneous (SC) x1; then pregabalin 150mg (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive placebo in the same dosing scheme.
  Other Names: Pregabalin/Placebo
  Arms: Pregabalin, then Placebo
Drug: Placebo — During the first chemotherapy cycle, the patient will receive placebo (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then placebo (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive pregabalin in the same dosing scheme.
  Other Names: Placebo/Pregabalin
  Arms: Placebo, then Pregabalin

SUMMARY:
Purpose:

To evaluate the preventative effects of pregabalin on pegfilgrastim-induced bone pain in cycle 1. Because granulocyte colony stimulating factor (G-CSF) receptors are found at nerve endings which modulate the pain signal, blocking this with pregabalin is theorized to prevent the occurrence of this adverse effect.

Participants:

Patients will be at least 18 years of age with either a diagnosis of a non-myeloid hematologic malignancy scheduled to initiate a cycle of chemotherapy that requires prophylactic use of a G-CSF, or with a diagnosis of breast cancer scheduled to initiate dose-dense doxorubicin/cyclophosphamide chemotherapy or docetaxel/cyclophosphamide that requires prophylactic use of a G-CSF.

Procedures (methods):

This is a randomized (1:1), single center, placebo-controlled, double blind, crossover phase II study. The primary objective is to compare the proportion of patients who have an increase in pain score of ≥3 from baseline in cycle 1 between Arm A (pregabalin) and Arm B (placebo). In consultation with the treating physician, the PI will determine what day pegfilgrastim will be initiated in each eligible, consented patient. Pregabalin or placebo will begin 4 days prior to pegfilgrastim administration, and continue for 7 additional days starting the day of pegfilgrastim administration.

DETAILED DESCRIPTION:
**Study Synopsis**

This is a randomized, double-blind, placebo-controlled, single center, crossover phase II clinical trial investigating the prophylactic analgesic effects of pregabalin (Lyrica®) during the first two cycles of chemotherapy in cancer patients receiving pegfilgrastim (Neulasta®). The investigators have restricted enrollment in this trial to breast cancer patients and those with hematological malignancies, who require pegfilgrastim prophylactically. Pegfilgrastim is associated with bone pain (which can be severe) when used in these populations.

In this study 60 patients are randomized to Arm A (pregabalin in cycle 1; placebo in cycle 2) or Arm B (placebo in cycle 1; pregabalin in cycle 2). The primary objective is to compare the proportion of patients who have an increase in pain score of ≥3 from baseline through the end of study medication in cycle 1 between Arm A (pregabalin) and Arm B (placebo).

A secondary objective is to compare of the proportion of patients with an increase in pain score of ≥3 from baseline between pregabalin and placebo across the 2 cycles. Other outcomes evaluated are the safety of this combination, the proportion of patients with an increase in bone/joint pain score of ≥3 from baseline, the proportion of patients with severe pain, the maximum change in pain score, and time to and number of days of rescue (breakthrough) analgesics.

For measuring pain, the investigators will rely on a validated 10-point numerical pain scale that patients will complete prior to initiation of pregabalin in each cycle, and for 7 days starting the day of pegfilgrastim administration in each cycle.

Pegfilgrastim is a pegylated form of granulocyte colony-stimulating factor (G-CSF) which is FDA approved to decrease the duration of neutropenia, thus the incidence of infection, by stimulating granulocyte production in patients receiving myelosuppressive chemotherapy associated with a significant risk of febrile neutropenia. As a long-acting product, this pegylated version is administered once per chemotherapy cycle, 24-72 hours after chemotherapy is complete.

Bone and skeletal pain due to pegfilgrastim have been reported in early clinical trials at rates of 22-33%, with sites of pain commonly noted in the lower back, posterior iliac crest and sternum. However more recent studies have found incidences as high as 59-71% with 27% experiencing severe pain (pain greater than 5 on a 10-point scale). Notably, Kirshner and colleagues conducted a phase III randomized trial evaluating the non-steroidal anti-inflammatory (NSAID) naproxen for the prevention of pegfilgrastim-related bone pain in patients with nonmyeloid cancer. Patients completed questionnaires at home documenting any new bone or joint pain post pegfilgrastim. The majority enrolled (68%) had breast cancer, and 7% had hematological malignancies. In this study of 510 patients, (257 on naproxen and 253 on placebo), the overall pain incidence was 71.3% (27% severe) in the placebo group and 61.1 % (19.2% severe) in the naproxen group. While naproxen significantly reduced the incidence of all and severe bone pain, and reduced the duration of bone pain (from 2.4 to 1.9 days), the authors concluded that novel preventive strategies are needed given the high incidence of bone pain even when naproxen is used for treatment.

The average onset of bone pain is 4 days after initiation of pegfilgrastim and with a duration of between 2-3 consecutive days. Because patients get multiple cycles of chemotherapy every 14-28 days, these repeated episodes of bone pain can significantly hinder quality of life. In the case where pegfilgrastim is withheld because of severe bone pain, chemotherapy dose-intensity and schedule often cannot be maintained threatening efficacy in addition to an increased potential for infectious complications.

Bone pain secondary to pegfilgrastim is usually treated with NSAIDs such as ibuprofen or naproxen, or opioids. Opioids are often preferred over NSAIDs because patients may be thrombocytopenic and at risk for gastrointestinal bleeding, and NSAIDs increase the risk of both of these adverse events. In addition, NSAIDs have an antipyretic property which is problematic in neutropenic patients. Their use can mask febrile neutropenia, which could mean an important sign of infection is missed in immunocompromised hosts. Because there are no established predictive factors for development of bone pain, nearly all patients who get pegfilgrastim receive a prescription for opioids in case they experience pain. Patients do not take pain medications to prevent the pain, but instead generally wait until they experience pain before starting these analgesics. In general, pain is more difficult to control once it has started, thus a prophylactic strategy may be more advantageous. To avoid any impact on the dose and/or schedule of chemotherapy, it would be optimal to prevent bone pain occurring after administration of pegfilgrastim, rather than advising the patient to treat this pain if/when it happens.

Primary Objective

Compare the proportion of patients who have an increase in pain score of ≥ 3 from baseline through the end of study medication in cycle 1 between Arm A and Arm B

Secondary Objectives

* Compare the proportion of patients who have an increase in pain score of ≥ 3 from baseline between pregabalin and placebo across the 2 cycles
* Compare the proportion of patients who have an increase in bone/joint pain score of ≥ 3 from baseline through the end of study medication in cycle 1 between Arm A and Arm B
* Compare the number of days of breakthrough analgesic use between pregabalin and placebo within cycle 1 and across the 2 cycles
* Compare the proportion of patients with severe pain between pregabalin and placebo within cycle 1 and across the 2 cycles
* Compare the maximum change in pain score from baseline between pregabalin and placebo within cycle 1 and across the 2 cycles
* Compare the maximum neuropathic pain score between pregabalin and placebo within cycle 1 and across the 2 cycles
* Describe the safety (assessed via NCI CTCAE v4) of pregabalin when used in the prevention of bone pain secondary to pegfilgrastim

Exploratory Objective

* Compare pain measures between pregabalin and placebo in the breast cancer and hematological malignancy subgroups separately within cycle 1 and across the 2 cycles
* Compare the time to first breakthrough analgesic use between pregabalin and placebo during cycle 1

Primary Endpoint

Pain score is based on a 10-point numerical scale (see section 11.1) for pain as documented at baseline (at screening for cycle 1 and day 1 of study medication prior to cycle 2) and on patient log (see section 11.3) for 7 days starting the day of pegfilgrastim administration

Secondary/Exploratory Endpoints

* Bone/joint pain score is based on a 10-point numerical scale (see section 11.1) for pain as documented at baseline (at screening for cycle 1 and day 1 of study medication prior to cycle 2) and on patient log (see section 11.3) for 7 days starting the day of pegfilgrastim administration
* Severe pain will be measured using the 10-point numerical scale for pain (see section 11.1) as documented on the patient log (section 11.3; severe pain is defined as a score >5 on this scale, similar to Kirshner and colleagues3)
* A day of breakthrough analgesic use is defined as any day in which patient increases the dose of any pain medication compared to baseline, or the addition of a new pain medication as documented on patient log (see section 11.3); time to first breakthrough analgesic use is defined as the time in days from pegfilgrastim administration to the first day patient uses breakthrough analgesic
* Neuropathic pain is assessed via the Neuropathic Pain Scale (see section 11.2) as documented from phone calls twice during study medication administration post pegfilgrastim administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of a non-myeloid hematologic malignancy scheduled to initiate a cycle of chemotherapy that requires prophylactic use of a granulocyte colony-stimulating growth factor (based on the provider's discretion), provided the schedule of chemotherapy cycles allows the use of pegfilgrastim at a dose of 6 mg SC once per cycle OR Diagnosis of breast cancer scheduled to initiate dose-dense doxorubicin and cyclophosphamide (AC) chemotherapy or docetaxel and cyclophosphamide (TC) chemotherapy that requires prophylactic use of a granulocyte colony-stimulating growth factor, provided the schedule of chemotherapy cycles allows the use of pegfilgrastim, at a dose of 6 mg SC once per cycle; pegfilgrastim scheduled for 24 hours post chemotherapy.
* Schedule of chemotherapy and pegfilgrastim initiation can accommodate initiation of pregabalin 4 days prior to pegfilgrastim dose.
* Baseline pain scores <7 as measured via 10-point numerical scale for pain (see section 11.1); pain score and use of any non-opioid pain medication must be self-reported as stable (same dose and frequency) over the 7 days prior to screening; for opioids, patient must self-report the same dose and frequency over the 28 days prior to screening. Patients who are receiving peri-procedural short-acting analgesics will still be included as long as they are no longer receiving analgesics by D1 of chemotherapy.

Exclusion Criteria:

* A history of (within one month) or current pregabalin use.
* Baseline pain scores ≥7 as measured via 10-point numerical scale for pain (see section 11.1).
* Unwilling to discontinue use of antihistamines from 7 days prior to D1 of study medication.
* Creatinine clearance (CrCl) ≤60 ml/min (as measured via Cockcroft-Gault) based on serum creatinine measured as part of standard of care prior to administration of chemotherapy
* Women of childbearing potential must have a negative serum pregnancy test prior to initiating therapy (note, this test should be standard of care prior to administration of chemotherapy).
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator.
* Eligible and agrees to enroll into therapeutic trial ongoing at the Lineberger Comprehensive Cancer Center (LCCC) (i.e., the treatment trial will take precedence over LCCC1314).
* Currently receiving therapeutic doses of anticoagulants (ie, prophylactic use of anticoagulants is allowed) due to possibility of dizziness and falls while on pregabalin.
* Currently receiving aromatase inhibitors or agents targeted against Ph+ leukemias (i.e., imatinib, dasatinib, nilotinib, and ponatinib) or scheduled to start these drugs during cycle 1 of scheduled chemotherapy.
* Presence of bone metastases.
* History of angioedema.
* History of a seizure disorder.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benyam Muluneh, PharmD, CPP, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared and kept confidential.

REFERENCES:
- [Background] Amgen. Pegfilgrastim. Package Insert. Accessed June 9, 2013
- [Background] Kirshner J, Hickock J, Hofman M. Pegfilgrastim-induced bone pain: Incidence, risk factors, and management in a community practice. Comm Onc 4:455-459, 2007.
- [Background] Kirshner JJ, Heckler CE, Janelsins MC, Dakhil SR, Hopkins JO, Coles C, Morrow GR. Prevention of pegfilgrastim-induced bone pain: a phase III double-blind placebo-controlled randomized clinical trial of the university of rochester cancer center clinical community oncology program research base. J Clin Oncol. 2012 Jun 1;30(16):1974-9. doi: 10.1200/JCO.2011.37.8364. Epub 2012 Apr 16. PMID 22508813
- [Background] Kubista E, Glaspy J, Holmes FA, Green MD, Hackett J, Neumann T; Pegfilgrastim Study Group. Bone pain associated with once-per-cycle pegfilgrastim is similar to daily filgrastim in patients with breast cancer. Clin Breast Cancer. 2003 Feb;3(6):391-8. doi: 10.3816/cbc.2003.n.003. PMID 12636878
- [Background] Tassone DM, Boyce E, Guyer J, Nuzum D. Pregabalin: a novel gamma-aminobutyric acid analogue in the treatment of neuropathic pain, partial-onset seizures, and anxiety disorders. Clin Ther. 2007 Jan;29(1):26-48. doi: 10.1016/j.clinthera.2007.01.013. PMID 17379045
- See also: University of North Carolina (UNC) Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11/2015 through 07/2017.
Pre-assignment Details: Eleven subjects were screened and successfully consented to this trial. Of these, three subjects either had therapy alteration that led to their exclusion or left without study-related medication, thus 8 subjects were treated.
Groups:
- Pregabalin, Then Placebo: Pregabalin in cycle 1; placebo in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg BID for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Pregabalin: During the first chemotherapy cycle, the patient will receive pregabalin 75mg (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then pregabalin 150mg (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive placebo in the same dosing scheme.
- Placebo, Then Pregabalin: Placebo in cycle 1; pregabalin in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg BID for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Placebo: During the first chemotherapy cycle, the patient will receive placebo (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then placebo (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive pregabalin in the same dosing scheme.
Period: First Intervention
Arm/Group | Pregabalin, Then Placebo | Placebo, Then Pregabalin
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0
Period: Washout
Arm/Group | Pregabalin, Then Placebo | Placebo, Then Pregabalin
Started | 5 | 3
Completed | 4 | 3
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention
Arm/Group | Pregabalin, Then Placebo | Placebo, Then Pregabalin
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin, Then Placebo | Placebo, Then Pregabalin | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 46.2 [23 to 71] | 51.3 [33 to 62] | 48.1 [23 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 3 | 8
Serum creatinine (SCr) [Mean (Full Range); unit: mg/dL] | 0.7 [0.5 to 0.9] | 0.6 [0.6 to 0.7] | 0.7 [0.5 to 0.9]
Baseline pain score [Mean (Full Range); unit: units on a scale] — The ten-point numerical scale is scored as an integer from 0 to 10. Participants will use this scale to rate their pain (and separately bone/joint pain) with 0 signifying "no pain" and 10 signifying "the worst pain you can imagine." As such, higher values (approaching 10) signify worse outcomes.
  units on a scale | 0.8 [0 to 2] | 3.3 [2 to 6] | 1.8 [0 to 6]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 28.2 [20.1 to 32.0] | 24.3 [20.6 to 26.8] | 26.7 [20.1 to 32.0]
Body Surface Area (BSA) [Mean (Full Range); unit: m^2] | 1.89 [1.68 to 2.16] | 1.86 [1.82 to 1.91] | 1.88 [1.68 to 2.16]
Eastern Cooperative Oncology Group (ECOG) performance status [Mean (Full Range); unit: units on a scale] — Measure Description: A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  units on a scale | 0.4 [0 to 1] | 0.3 [0 to 1] | 0.4 [0 to 1]
Baseline neuropathic pain scale [Mean (Full Range); unit: units on a scale] — The ID-Pain scale (i.e. neuropathic pain scale) is a 6-item, participant-completed screening tool to help differentiate nociceptive and neuropathic pain.
  1. Did the pain feel like pins and needles?
  2. Did the pain feel hot/burning?
  3. Did the pain feel numb?
  4. Did the pain feel like electrical shocks?
  5. Is the pain made worse with the touch of clothing or bed sheets?
  6. Is the pain limited to your joints?
  A "yes" response to questions 1-5 are scored as 1; for question 6, is scored as -1. As such, higher scores (approaching 5) signify worse outcomes. Scale total range of -1 to 5.
  units on a scale | 0 [0 to 0] | 0.3 [0 to 1] | 0.1 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Have an Increase in Pain Score of ≥ 3 From Baseline Through the End of Study Medication in Cycle 1
Description: Compare the proportion of patients who have an increase in pain score of ≥ 3 from baseline through the end of study medication in cycle 1 between Arm A and Arm B.
  The ten-point numerical scale is scored from 0 to 10. They will use this scale to rate their pain (and separately bone/joint pain) with 0 signifying "no pain" and 10 signifying "the worst pain you can imagine."
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- First Intervention = Pregabalin: Pregabalin in cycle 1; placebo in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg twice a day (BID) for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Pregabalin: During the first chemotherapy cycle, the patient will receive pregabalin 75mg (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then pregabalin 150mg (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive placebo in the same dosing scheme.
- First Intervention = Placebo: Placebo in cycle 1; pregabalin in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg BID for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Placebo: During the first chemotherapy cycle, the patient will receive placebo (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then placebo (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive pregabalin in the same dosing scheme.
Arm/Group | First Intervention = Pregabalin | First Intervention = Placebo
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

2. Secondary Outcome: Proportion of Patients Who Have an Increase in Pain Score of ≥ 3 From Baseline Between Pregabalin and Placebo Across the 2 Cycles
Description: Compare the proportion of patients who have an increase in pain score of ≥ 3 from baseline between pregabalin and placebo across the 2 cycles.
  The ten-point numerical scale is scored from 0 to 10. They will use this scale to rate their pain (and separately bone/joint pain) with 0 signifying "no pain" and 10 signifying "the worst pain you can imagine."
Time Frame: Up to 12 weeks
Measure: Number; unit: proportion
Groups:
- First Intervention = Pregabalin; Second Intervention = Placebo: Pregabalin in cycle 1; placebo in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg BID for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Pregabalin: During the first chemotherapy cycle, the patient will receive pregabalin 75mg (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then pregabalin 150mg (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive placebo in the same dosing scheme.
- Second Intervention = Pregabalin: Placebo in cycle 1; pregabalin in cycle 2.
  Pregabalin or matching placebo will be administered at 75 mg BID for 4 days, to patients receiving pegfilgrastim for hematologic malignancies or breast cancer patients on myelosuppressive chemotherapy . Starting the day of pegfilgrastim, the dose of study medication will be increased to 150 mg PO BID provided the patient is tolerating the lower dose (ie, they are not experiencing any pregabalin associated toxicities >Grade 1). This will be determined by the research team on the day of pegfilgrastim administration.
  Placebo: During the first chemotherapy cycle, the patient will receive placebo (1 capsule) BID x 4 days before pegfilgrastim 6mg SC x1; then placebo (2 capsules) BID x 7 days. During the second chemotherapy cycle, the patient will receive pregabalin in the same dosing scheme.
Arm/Group | First Intervention = Pregabalin | Second Intervention = Placebo | First Intervention = Placebo | Second Intervention = Pregabalin
Number analyzed (Participants) | 5 | 4 | 3 | 3
proportion | 0 | 0.5 | 0 | 0.333

3. Secondary Outcome: Proportion of Patients Who Have an Increase in Bone/Joint Pain Score of ≥ 3 From Baseline Through the End of Study Medication in Cycle 1
Description: Compare the proportion of patients who have an increase in bone/joint pain score of ≥ 3 from baseline through the end of study medication in cycle 1 between Arm A and Arm B.
  The ten-point numerical scale is scored from 0 to 10. They will use this scale to rate their pain (and separately bone/joint pain) with 0 signifying "no pain" and 10 signifying "the worst pain you can imagine."
Time Frame: Up to 12 weeks
Measure: Number; unit: proportion
Arm/Group | First Intervention = Pregabalin | First Intervention = Placebo
Number analyzed (Participants) | 5 | 3
proportion | 0 | 0

4. Secondary Outcome: Number of Days of Breakthrough Analgesic Use Between Pregabalin and Placebo Across the 2 Cycles
Description: Compare the number of days of breakthrough analgesic use between pregabalin and placebo within cycle 1 and across the 2 cycles.
  The number of days of breakthrough analgesic use (i.e additional pain medication being required) is evaluated based on participant-provided medication logs kept during study treatment. If additional pain medication outside of their normal pain control regimen was reported, this day counts as 1. The total days for each patient are then reported, with a total range from zero to 14 (for patients with breast cancer) or zero to 21 (for patients with a lymphoma).
Time Frame: Up to 12 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | First Intervention = Pregabalin | Second Intervention = Placebo | First Intervention = Placebo | Second Intervention = Pregabalin
Number analyzed (Participants) | 5 | 4 | 3 | 3
days | 1.4 [0 to 5] | 3.25 [0 to 13] | 0.67 [0 to 1] | 0 [0 to 0]

5. Secondary Outcome: Proportion of Patients With Severe Pain Between Pregabalin and Placebo Across the 2 Cycles
Description: Compare the proportion of patients with severe pain between pregabalin and placebo within cycle 1 and across the 2 cycles.
  The ten-point numerical scale is scored from 0 to 10. They will use this scale to rate their pain (and separately bone/joint pain) with 0 signifying "no pain" and 10 signifying "the worst pain you can imagine."
Time Frame: Up to 12 weeks
Measure: Number; unit: proportion
Arm/Group | First Intervention = Pregabalin | Second Intervention = Placebo | First Intervention = Placebo | Second Intervention = Pregabalin
Number analyzed (Participants) | 5 | 4 | 3 | 3
proportion | 0.4 | 0.25 | 0.67 | 0

6. Secondary Outcome: Maximum Change in Pain Score From Baseline Between Pregabalin and Placebo Across the 2 Cycles
Description: Compare the maximum change in pain score from baseline between pregabalin and placebo within cycle 1 and across the 2 cycles.
  The ten-point numerical scale is scored from 0 to 10. They will use this scale to rate their pain (and separately bone/joint pain) with 0 signifying "no pain" and 10 signifying "the worst pain you can imagine." Each patient will be assessed regularly, including: before therapeutic intervention (i.e. at consent/screening), first day of chemotherapy administration (during cycles 1 & 2), 4 days after pegfilgrastim administration (during cycles 1 & 2), and 8 days after pegfilgrastim administration (during cycles 1 & 2).
Time Frame: Up to 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | First Intervention = Pregabalin | Second Intervention = Placebo | First Intervention = Placebo | Second Intervention = Pregabalin
Number analyzed (Participants) | 5 | 4 | 3 | 3
units on a scale | 0.4 [0 to 2] | 2 [0 to 4] | 0 [0 to 0] | 1.67 [0 to 5]

7. Secondary Outcome: Maximum Neuropathic Pain Score Between Pregabalin and Placebo Across the 2 Cycles
Description: Compare the maximum neuropathic pain score between pregabalin and placebo within cycle 1 and across the 2 cycles.
  The "ID Pain" scale (also know as the "Identify Pain" scale) is a 6-item, participant-completed screening tool designed to help differentiate nociceptive and neuropathic pain. This pain score also helps to evaluate the presence/absence of neuropathic pain at a given point of time.
  1. Did the pain feel like pins and needles?
  2. Did the pain feel hot/burning?
  3. Did the pain feel numb?
  4. Did the pain feel like electrical shocks?
  5. Is the pain made worse with the touch of clothing or bed sheets?
  6. Is the pain limited to your joints?
  A "yes" response to questions 1-5 are scored as 1; for question 6, a "yes" is scored as -1. As such, higher scores (approaching 5) signify worse outcomes. The scale's total range for a patient is -1 to 5.
Time Frame: Up to 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | First Intervention = Pregabalin | Second Intervention = Placebo | First Intervention = Placebo | Second Intervention = Pregabalin
Number analyzed (Participants) | 5 | 4 | 3 | 3
units on a scale | 0.2 [0 to 1] | 0.5 [0 to 2] | 0 [0 to 0] | 0.33 [0 to 1]

8. Secondary Outcome: Number of Subjects That Experienced a Grade 2 or Higher Adverse Events When Taking Pregabalin
Description: CTCAE The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | First Intervention = Pregabalin | Second Intervention = Pregabalin
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During the first two cycles of therapy (roughly 12 weeks from initiation of therapy), or during a total of 24 weeks. Each patient will be assessed regularly for the development of any toxicity, including: before therapeutic intervention (i.e. at consent/screening), first day of chemotherapy administration (during cycles 1 & 2), 4 days after pegfilgrastim administration (during cycles 1 & 2), and 8 days after pegfilgrastim administration (during cycles 1 & 2).
Arm/Group | First Intervention = Pregabalin | Second Intervention = Placebo | First Intervention = Placebo | Second Intervention = Pregabalin
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Intervention = Pregabalin (N=5) | Second Intervention = Placebo (N=4) | First Intervention = Placebo (N=3) | Second Intervention = Pregabalin (N=3)
Fatigue (General disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drowsiness/Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
We were unable to achieve the target number of subject participants (target n=60; accrual n=11) needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03407430/Prot_SAP_004.pdf